CLINICAL TRIAL: NCT04684563
Title: Phase I Trial of huCART19-IL18 Cells in Patients With Relapsed or Refractory CD19+ Cancers
Brief Title: huCART19-IL18 in CD19+ Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: BlueWhale Bio (Cohort D only) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15420; IRB# 844955
Record Dates: First submitted 2020-12-11; First posted 2020-12-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; Non-hodgkin Lymphoma; Acute Lymphoblastic Leukemia
Keywords: CLL; NHL; CAR-T cells
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Cohort A: NHL Dose Level 1a (DL1a) (Experimental): 3x10^6 huCART19-IL18 cells administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level -1 (DL-1) (Experimental): 7x10^5 huCART19-IL18 cells administered as a single intravenous (IV) infusion or slow IV push; This dose level will only be explored if at least one DLT is observed at Dose Level 1a.
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level 1b (DL1b) (Experimental): 3x10^6 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level 2 (DL2) (Experimental): 7x10^6 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level 3 (DL3) (Experimental): 3x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level 4 (DL4) (Experimental): 7x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort A: NHL Dose Level 5 (DL5) (Experimental): 3x10^8 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort B: CLL Dose Level 1b (DL1b) (Experimental): 3x10^6 huCART19-IL18 cells administered as a single intravenous (IV) infusion or slow IV push; This dose level will only be explored if at least one DLT is observed at Dose Level 2.
  Interventions: Biological: huCART19-IL18
- Cohort B: CLL Dose Level 2 (DL2) (Experimental): 7x10^6 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort B: CLL Dose Level 3 (DL3) (Experimental): 3x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort B: CLL Dose Level 4 (DL4) (Experimental): 7x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort B: CLL Dose Level 5 (DL5) (Experimental): 3x10^8 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort C: ALL Dose Level 1b (DL1b) (Experimental): 3x10^6 huCART19-IL18 cells administered as a single intravenous (IV) infusion or slow IV push; This dose level will only be explored if at least one DLT is observed at Dose Level 2.
  Interventions: Biological: huCART19-IL18
- Cohort C: ALL Dose Level 2 (DL2) (Experimental): 7x10^6 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort C: ALL Dose Level 3 (DL3) (Experimental): 3x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort C: ALL Dose Level 4 (DL4) (Experimental): 7x10^7 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort C: ALL Dose Level 5 (DL5) (Experimental): 3x10^8 huCART19-IL18 cells following lymphodepleting chemotherapy administered as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort D: NHL (Experimental): 7x10^6 huCART19-IL18 as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18
- Cohort D: ALL (Experimental): 7x10^6 huCART19-IL18 as a single intravenous (IV) infusion or slow IV push
  Interventions: Biological: huCART19-IL18

INTERVENTIONS:
Biological: huCART19-IL18 — autologous Chimeric Antigen Receptor (CAR) T cells directed against the human CD19 antigen that also express human Interleukin 18 (IL-18)

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of huCART19-IL18 cells in patients with relapsed or refractory CD19+ cancers.

DETAILED DESCRIPTION:
This is a Phase I study to assess the safety, tolerability, manufacturing feasibility, pharmacokinetics, and preliminary efficacy of huCART19-IL18 cells in patients with CD19+ cancers. The study will take place in two parts: an initial Dose-Finding Phase and an Expansion Phase. In the dose-finding phase, the maximum tolerated dose will be determined using a Bayesian Optimal Interval (BOIN) design within each of the following disease-specific cohorts:

* Cohort A: Non-Hodgkin Lymphoma (Active, Not Recruiting)
* Cohort B: Chronic Lymphocytic Leukemia (Active, Not Recruiting)
* Cohort C: Acute Lymphoblastic Leukemia (Active, Not Recruiting)
* Cohort D (Expansion Phase): Non Hodgkin Lymphoma and Acute Lymphoblastic Leukemia (Active, Not Recruiting) will evaluate changes to cell activation method in the huCART19-IL18 manufacturing process using the recommended dose for expansion (RDE) arising out of the dose-finding phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Documentation of CD19 expression on malignant cells by flow cytometry/IHC from a CLIA certified laboratory

   NHL Patients: Within 6 months of physician-investigator confirmation of eligibility as long as there has been no intervening CD19 directed therapy since expression confirmed. Results outside of this window may be used, if there is no accessible tumor site and the subject did not receive intervening CD19 directed therapy since CD19 expression was confirmed.

   CLL and ALL Patients: At time of most recent relapse. If the subject has subsequently received CD19-directed therapy since this result was obtained, repeating testing must be performed to determine eligibility.
3. Patients with relapsed disease after prior allogeneic SCT must meet the following criteria:

   a. Have no active GVHD and require no immunosuppression b. Are more than 6 months from transplant at the time of physician-investigator confirmation of eligibility
4. Adequate organ function defined as:

   a. Creatinine ≤ 1.6 mg/dl b. ALT/AST ≤ 3x upper limit of normal range c. Direct bilirubin ≤ 2.0 mg/dl, unless the subject has Gilbert's syndrome (≤3.0 mg/dl) d. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air e. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
5. Evidence of active disease within 12 weeks of physician-investigator confirmation of eligibility. .
6. Male or female age ≥ 18 years.
7. ECOG Performance Status that is either 0 or 1.
8. Subjects of reproductive potential must agree to use acceptable birth control methods.
9. Disease-specific criteria:

NHL Patients (Cohorts A and D):

i. Patients with any of the following diagnoses: Diffuse Large B-cell Lymphoma not otherwise specified (DLBCL NOS), germinal center or activated B-cell types;Primary Cutaneous DLBCL; Primary Mediastinal (thymic) Large B-cell Lymphoma; ALK+ Anaplastic Large B-cell Lymphoma; High-Grade B-cell Lymphoma with MYC and BCL2 and/or BCL6 rearrangements (i.e., "Double or Triple Hit"); High-grade B-cell Lymphoma, NOS; T-cell Rich B-cell Lymphoma; Transformed Follicular Lymphoma; or any aggressive B-cell lymphoma arising from indolent lymphoma.

1. Patients must have either relapsed after, or be ineligible for, prior CAR T cell therapy, and meet one of the following criteria:

1. Relapsed/refractory disease after at least 2 prior lines of appropriate therapy; OR
2. Relapsed/refractory disease after autologous SCT; OR
3. Relapsed/refractory disease after allogeneic SCT. ii. Follicular lymphoma

   1. Patients must have either relapsed after, or be ineligible for, prior commercial CAR T cell therapy; AND
   2. Received at least 2 prior lines of appropriate therapy (not including single agent monoclonal antibody therapy) and progressed within 2 years after second or higher line of therapy.

iii. Mantle cell lymphoma

1. Patients must have either failed standard of care CAR T cell therapy (e.g., Tecartus™, etc) or other investigational CAR T cell product, OR be ineligible for standard of care Tecartus™; and
2. Patients must also meet one of the following criteria:

   1. Relapsed/refractory disease after at least 2 prior lines of appropriate therapy, including a BTK inhibitor. Single-agent monoclonal antibody therapy does not count towards prior lines of therapy; OR
   2. Relapsed/refractory disease after prior autologous SCT; OR
   3. Relapsed/refractory disease after prior allogeneic SCT.

CLL Patients (Cohort B):

i. Chronic Lymphocytic Leukemia

1. Patients with relapsed/refractory disease after at least 2 prior lines of appropriate therapy; AND
2. Patients must have previously received or be intolerant to an approved BTK inhibitor and venetoclax, unless a BTK inhibitor or venetoclax is contraindicated.

ii. Large cell transformation of CLL (Richter's Transformation)

1. Patients must be primary refractory or received at least 1 prior line of treatment for Richter's Transformation.

c. ALL Patients (Cohorts C and D): i. Patients with b-cell acute lymphoblastic leukemia. Note: Chronic myeloid leukemia (CML) lymphoid blast crisis is considered a sub-type of relapsed B-ALL, thus will be encompassed in our definition of B-ALL throughout; AND ii. Patients with 2nd or greater relapse or refractory disease as defined by one of the following criteria:

1. Recurrent disease in the blood or bone marrow identified morphologically, by IHC or flow; OR
2. Isolated CNS disease. Note: Patients with prior/current history of CNS3 disease will only be eligible for treatment if the CNS disease is responsive to therapy; OR
3. Recurrent extramedullary disease at other (non-CNS) sites if disease response can be assessed radiographically. Note: Patients with recurrent extramedullary disease do not need to have detectable blood or bone marrow involvement; OR
4. Any relapse after allogeneic SCT; OR
5. Patients with refractory disease as defined by one of the following:

   1. Failure to achieve remission (<5% bone marrow blasts or ongoing extramedullary or CNS disease) after 2 cycles of induction chemotherapy; OR
   2. Patients that achieve remission but remain MRD+ after ≥2 cycles of induction chemotherapy.

Exclusion Criteria:

1. Active hepatitis B, active hepatitis C, or other active, uncontrolled infection.
2. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
3. Clinically apparent arrhythmia or arrhythmias that are not stable on medical management within two weeks of physician-investigator confirmation of eligibility.
4. Active acute or chronic GVHD requiring systemic therapy.
5. Dependence on systemic steroids or immunosuppressant medications. For additional details regarding use of steroid and immunosuppressant medications.
6. RETIRED WITH PROTOCOL AMENDMENT V7
7. Receipt of prior huCART19 therapy.
8. CNS disease as defined by disease-cohort as follows:

   1. NHL/CLL Patients: Active CNS disease. Note: Patients with a history of CNS involvement that was successfully treated are eligible. A CNS evaluation is only required for eligibility if a subject is experiencing signs/symptoms of CNS involvement.
   2. ALL Patients: CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
9. Pregnant or nursing (lactating) women.
10. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to their cancer or previous cancer treatment.
11. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2036-05 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | Up to 15 years post-huCART19-IL18 infusion
  Cohorts A-C: Type, frequency and severity of adverse events as assessed by CTCAE V5.0. Each disease-specific cohort will be analyzed separately.
Occurrence of dose-limiting toxicities (DLTs) | 28 days post-huCART19-IL18 infusion
  Cohorts A-C: Unacceptable toxicity as defined by the protocol. DLTs will be evaluated separately by each disease-specific cohort.
Determination of Maximum Tolerated Dose (MTD) | 28 days post-huCART19-IL18 infusion
  Cohorts A-C: Selected based on an isotonic regression model. The MTD will be established separately by disease-specific cohort.
Determination of a recommended dose for expansion (RDE) | 3 months post-huCART19-IL18 infusion
  Cohorts A-C: Evaluated by Cohort/dose level using a multi-criteria decision analysis.
Proportion of manufactured products that meet the product release criteria | 3 months
  Cohort D: Calculated based on the proportion of subjects with huCART19-IL18 products that fail to meet the product release criteria, out of the number of subjects in whom manufacturing was attempted.
Proportion of manufactured products that meet the assigned dose | 3 months
  Cohort D: Calculated based on the proportion of subjects with huCART19-IL18 products that fail to meet the assigned dose, out of the number of subjects in whom manufacturing was attempted.

SECONDARY OUTCOMES:
Proportion of manufacturing products that meet the product release criteria | 3 months
  Cohorts A-C: Calculated based on the proportion of subjects with huCART19-IL18 products that fail to meet the product release criteria, out of the number of subjects in whom manufacturing was attempted. Will be evaluated separately by each disease-specific cohort.
Proportion of manufactured products that meet the assigned dose | 3 months
  Cohorts A-C: Calculated based on the proportion of subjects with huCART19-IL18 products that fail to meet the assigned dose, out of the number of subjects in whom manufacturing was attempted. Will be evaluated separately by each disease-specific cohort.
Incidence of Treatment-Emergent Adverse Events | 3 months
  Cohort D: Type, frequency and severity of adverse events as assessed by CTCAE V5.0.
Overall Response Rate (ORR) | 3 months post-huCART19-IL18 infusion
  NHL and CLL Patients: The proportion of subjects with CR or PR at Month 3 as compared to baseline.
Overall Response Rate (ORR) | 1 month post-huCART19-IL18 infusion
  ALL Patients: The proportion of subjects with CR/CRi/CR(MRD-) at Day 28 as compared to baseline
Best Overall Response (BOR) | 12 months post-huCART19-IL18 infusion
  NHL and CLL Patients: The proportion of subjects with a best overall disease response of CR or PR between Month 3 and Month 12, and prior to the start of new anticancer therapy.
Best Overall Response (BOR) | 6 months post-huCART19-IL18 infusion
  ALL Patients: The proportion of subjects with CR/CRi/CR(MRD-) by Month 6, and prior to the start of new anticancer therapy.
Duration of Response (DOR) | Up to 15 years post-huCART19-IL18 infusion
  NHL and CLL Patients: Duration from the date when CR/PR is first met at/after Month 3, to the date of relapse, death, or receipt of new anticancer therapy.
Duration of Remission (DOR) | Up to 15 years post-huCART19-IL18 infusion
  ALL Patients: Duration from the date when CR/CRi/CR(MRD-) is first met to the date of relapse, death or receipt of new anticancer therapy
Progression-Free Survival (PFS) | 12 monthsUp to 15 years post-huCART19-IL18 infusion
  NHL and CLL Patients: Duration of time from the huCART19-IL18 infusion to the date of the disease progression/relapse, death or receipt of new anticancer therapy
Event-Free Survival (EFS) | Up to 15 years post-huCART19-IL18 infusion
  ALL Patients: Duration of time from the huCART19-IL18 infusion to the date of relapse/treatment failure, death or receipt of new anticancer therapy.
Overall Survival (OS) | Up to 15 years post-huCART19-IL18 infusion
  Duration of time from the huCART19-IL18 infusion to the date of death, for any reason
Characterize low level disease and B cell assessment in response to huCART19-IL18 cells by Flow Cytometry | 12 months
  Polychromatic flow cytometry-based assessment of leukemia and B cells, extent and duration of leukemic response
Characterize low level disease and B cell assessment in response to huCART19-IL18 cells by Next Gen Sequencing | 12 months
  Presence or absence of malignant B cells by Next-Generation Immunoglobulin heavy chain Sequencing (NGIS)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svoboda J, Landsburg DJ, Gerson J, Nasta SD, Barta SK, Chong EA, Cook M, Frey NV, Shea J, Cervini A, Marshall A, Four M, Davis MM, Jadlowsky JK, Chew A, Pequignot E, Gonzalez V, Noll JH, Paruzzo L, Rojas-Levine J, Plesa G, Scholler J, Siegel DL, Levine BL, Porter DL, Ghassemi S, Ruella M, Rech A, Leskowitz RM, Fraietta JA, Hwang WT, Hexner E, Schuster SJ, June CH. Enhanced CAR T-Cell Therapy for Lymphoma after Previous Failure. N Engl J Med. 2025 May 8;392(18):1824-1835. doi: 10.1056/NEJMoa2408771. PMID 40334157